CLINICAL TRIAL: NCT06509152
Title: Theory of Mind-based Social Competence Group Intervention (ToM-SCGI) in Children With Autism Spectrum Disorder: a Randomized Controlled Trial
Brief Title: Theory of Mind-based Social Competence Group Intervention
Acronym: ToM-SCGI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B-BR-112-082
Record Dates: First submitted 2024-06-17; First posted 2024-07-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: theory of mind; social competence; randomized, controlled trial; group intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ToM-SCGI-12 (Experimental): The ToM-SCGI-12 is designed as a 12-week group intervention, with 60-minute sessions held weekly and led by trained therapists. Each group consists of 3 to 6 children with ASD, assigned based on assessments of children's age, verbal IQ, theory of mind abilities, and social skills. Caregivers can observe the children's performance in the group and document the group's themes and contents using observation and feedback forms. Caregiver meetings are conducted in the 6th and 12th weeks of the intervention to discuss the children's progress, enhance caregivers' interaction skills, and motivate continued practice at home. After the intervention concludes, caregivers' feedback is also collected through questionnaires to emphasize the role of family in the intervention.
  Interventions: Behavioral: Theory of mind-based social competence group intervention
- ToM-SCGI-6 (Active Comparator): The ToM-SCGI-6 is designed as a 6-week group intervention, with two 60-minute sessions held weekly and led by trained therapists. Each group consists of 3 to 6 children with ASD, assigned based on assessments of children's age, verbal IQ, theory of mind abilities, and social skills. Caregivers can observe the children's performance in the group and document the group's themes and contents using observation and feedback forms. Caregiver meetings are conducted in the 6th and 12th weeks of the intervention to discuss the children's progress, enhance caregivers' interaction skills, and motivate continued practice at home. After the intervention concludes, caregivers' feedback is also collected through questionnaires to emphasize the role of family in the intervention.
  Interventions: Behavioral: Theory of mind-based social competence group intervention
- Control group (No Intervention): The control group participated in conventional occupational therapy that did not focus on theory of mind or social competence. The duration and length of the intervention were the same as those of the experimental group.

INTERVENTIONS:
Behavioral: Theory of mind-based social competence group intervention — The ToM-SCGI is designed as a group intervention, with 60-minute sessions held weekly, either once or twice, and led by trained therapists. Two caregiver meetings are conducted in the middle and end of the interventions.
  The intervention process for each session is as follows:
  1. Warm-up Activities(5-10 minutes): review the previous group session and prepare for the current group activities.
  2. Theory of Mind Instruction(10-15 minutes): based on the developmental stage of the children's theory of mind, using thought bubbles to teach corresponding elements of theory of mind development.
  3. Social Skills Group Games(30-35 minutes): design social scenario-based group games that allow children to practice applying the acquired theory of mind abilities into expressions and applications of theory of mind and social competence.
  4. Summary(5-10 minutes): summarize the children's performance in the group and assign homework.
  Arms: ToM-SCGI-12; ToM-SCGI-6

SUMMARY:
This clinical study introduces a novel intervention, the Theory of Mind-Based Social Competence Group Intervention (ToM-SCGI), designed to improve theory of mind and social competence in children with autism spectrum disorder (ASD). Investigators hypothesize that the ToM-SCGI, which focuses on enhancing the ability to understand others' thoughts and feelings-known as "theory of mind"-will positively impact children's theory of mind abilities, application of these abilities, and overall social competence.

In a carefully structured randomized controlled trial (RCT), investigators aim to validate the effectiveness of the ToM-SCGI. Additionally, investigators will examine if a child's verbal IQ and social interaction style can influence the effectiveness of the ToM-SCGI. Through three comprehensive phases-developing and piloting the intervention, conducting the RCT, and examining the mediation and moderation effects-investigators expect that the ToM-SCGI will provide lasting benefits in the social development of children with ASD.

DETAILED DESCRIPTION:
This study is a single-blind RCT aiming to enroll 120 pairs of participants, comprising 120 children with ASD and caregivers. The participants will be equally divided into two experimental groups and a control group, with 40 pairs each. The experimental groups will participate in the Theory of Mind-Based Social Competence Group Intervention (ToM-SCGI) focusing on theory of mind and social competence, while the control group will engage in regular occupational therapy without a specific focus on theory of mind or social competence. One experimental group will receive the intervention once a week for 12 weeks, while the other will receive it twice a week for 6 weeks.

The study consists of four assessments: T0 screening, T1 pre-intervention, T2 post-intervention, and T3 follow-up three months later. The T0 assessment is conducted to screen and confirm eligibility. Randomization and allocation concealment are managed independently by a researcher not involved in the study, using Random Allocation Software 2.0. Randomly generated numbers and group assignments are placed in consecutively numbered, opaque, sealed envelopes. Once a child and caregiver provide consent and eligibility is confirmed, the envelopes are opened sequentially to assign participants to one of the experimental and control groups.

The T1 assessment establishes baseline data for efficacy evaluations before the interventions. All groups then undergo the respective interventions. The T2 assessment, conducted within one week after completing the interventions, serves as the post-intervention measure. The final T3 follow-up assessment takes place three months after the intervention ends, to evaluate long-term effects.

ELIGIBILITY:
Inclusion Criteria:

1. chronological age between 3 and 10 years;
2. diagnosed with Autism Spectrum Disorder (ASD), Autism, Asperger's Syndrome, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS) according to DSM-5 or the International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) criteria by a trained psychiatrist or pediatrician;
3. absence of additional neurological or psychiatric conditions;
4. a T-score of 60 or higher on the Social Responsiveness Scale-Second Edition (SRS-2) and a score of 30 or higher on the Childhood Autism Rating Scale™, Second Edition (CARS™2);
5. a Verbedal Comprehension Index (VCI) score of 70 or higher on the Wechsler Preschool and Primary Scale of Intelligence IV (WPPSI-IV) or the Wechsler Intelligence Scale for Children IV (WISC-IV).

Exclusion Criteria:

1. inability to follow instructions or complete the entire assessment process;
2. symptoms related to organic brain dysfunction (e.g., epilepsy);
3. uncorrectable auditory or visual impairments.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Observational Social Competence Assessment, OSCA | Up to 1 week before the intervention, up to 1 week after completing the intervention, and 3 months after completing the intervention.
  This study will utilize the OSCA to assess children's social competencies. The OSCA is a semi-structured assessment tool designed to evaluate the social competencies of children with Autism Spectrum Disorder (ASD) aged 3 to 12, and it can also measure the effectiveness of interventions.
Theory of Mind Assessment, ToMA | Up to 1 week before the intervention, up to 1 week after completing the intervention, and 3 months after completing the intervention.
  ToMA will be used to evaluate children's theory of mind capabilities. ToMA was based on the multidimensional framework of theory of mind. ToMA consists of 26 items that comprehensively cover cognitive and affective dimensions of theory of mind development for children aged 3 to 12. It spans three developmental stages: early, basic, and advanced, assessing elements such as emotional recognition, differing desires, basic false beliefs about unexpected contents and locations, hidden emotions, second-order false beliefs, lying, white lies, sarcasm, faux pas, and third-order false beliefs. The assessment is designed as a series of linked cartoon storybooks presented on a computer, integrating developmental elements into natural contexts to make the assessment interactive, engaging, and captivating for children, thereby maintaining their focus throughout the testing process.
Theory of Mind Task Battery, ToMTB | Up to 1 week before the intervention, up to 1 week after completing the intervention, and 3 months after completing the intervention.
  Children's theory of mind capabilities will be assessed using the ToMTB. Suitable for ages 3 to 12, ToMTB consists of 9 subtests with a total of 15 items. The assessment is conducted in a one-on-one setting where scenarios are presented in a storybook format, allowing children to respond either through gestures or verbally. The subtests are arranged in increasing order of difficulty and include recognition questions, confirmation questions, and control questions. Control questions aim to exclude the effects of attention, memory, and verbal comprehension and are not included in the overall score. The ToMTB takes about 20 minutes to complete and is validated for high internal consistency and test-retest reliability.
Theory of Mind Inventory-Second Edition, ToMI-2 | Up to 1 week before the intervention, up to 1 week after completing the intervention, and 3 months after completing the intervention.
  ToMI-2 will be utilized to assess children's theory of mind performance. ToMI-2 primarily consists of a caregiver-completed questionnaire that provides insights into children's naturalistic behaviors. The inventory features 60 questions. Scoring is done on a continuous scale, with caregivers marking a vertical line along a 20 cm line that ranges from 'completely disagree' to 'completely agree', to indicate the degree of a child's theory of mind performance.
Vineland Adaptive Behavior Scales, Third Edition, VABS-3 | Up to 1 week before the intervention, up to 1 week after completing the intervention, and 3 months after completing the intervention.
  VABS-3 will be employed to assess children's everyday social adaptation behaviors. The VABS-3 is a semi-structured interview questionnaire filled out by primary caregivers, applicable to children aged 3 to 12 years. The overall composite standard scores of the scale provide a comprehensive assessment of a child's personal and social competencies. The VABS-3 Socialization domain provides standard scores, percentile ranks, adaptive levels, and age-equivalent scores for a child's adaptive behaviors in social areas and subdomains, as well as a strengths and weaknesses analysis of adaptive behavior performances.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Lin Chen, Ph.D, Principal Investigator — Nattional Cheng Kung University

IPD SHARING:
Plan to Share IPD: No